CLINICAL TRIAL: NCT01621919
Title: Concentration of S-1 Metabolites in Tear and Plasma and Correlation With Its Side Effects in Patients Receiving S-1 Adjuvant Chemotherapy
Brief Title: Concentration of S-1 Metabolites in Tear and Plasma of Patients Receiving TS-1
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Namju Kim, Professor for clinical department, Seoul National University Bundang Hospital
Other Study IDs: TITAP
Record Dates: First submitted 2012-06-14; First posted 2012-06-18 (Estimated); Last update posted 2012-06-18 (Estimated); Status verified 2012-06

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasma tears
Oversight: Data Monitoring Committee: No

SUMMARY:
S-1 has been also shown to be an effective drug for palliative chemotherapy in Eastern and Western GC patients. Recently, some case and small-sized studies have been reported on lacrimal drainage obstruction(LDO)caused by S-1.Suggested mechanism of LDO involves direct secretion of S-1 into the tear; thus the concentration of S-1 metabolite in tear is expected to be high in patients who developed LDO than in patients without LDO. We investigate the concentration of S-1 and its metabolites in tear and plasma and find out its correlation with side effects such as LDO. These results will also help us identify patients who are at high risk of developing S-1-associated side effects.

DETAILED DESCRIPTION:
1. S-1 metabolites concentration in plasma

   1. factors affecting plasma concentration

      * surgery subtype
      * serum creatinine
   2. systemic adverse effects of S-1 and its correlation with plasma S-1 metabolites concentration

      * enteritis
      * fatigue
2. S-1 metabolites concentration in tears

   1. correlation of tear concentration with plasma concentration
   2. lacrimal drainage obstruction caused by S-1 administration, and its correlation with tear S-1 metabolites concentration
   3. lacrimal drainage obstruction caused by S-1 administration, and its correlation with plasma S-1 metabolites concentration

ELIGIBILITY:
Inclusion Criteria:

* Patients who received radical surgery for gastric cancer
* Patients who receiving S-1 adjuvant chemotherapy
* Patients who administrated S-1 for more than 7 days

Exclusion Criteria:

* who using eyedrop medication
* who has dry eye that tear cannot be sampled

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who receiving S-1 as an adjuvant chemotherapy after radial surgery for gastric cancer
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2010-12; Primary Completion 2012-12 (Estimated); Study Completion 2013-05 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Keun-Wook Lee, MD, Study Director — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea